CLINICAL TRIAL: NCT00139893
Title: A Randomized, Open-label, Two-way Crossover Trial to Determine the Pharmacokinetics of Metoclopramide When Administered as the Orally Disintegrating Tablet Compared to Reglan® Tablets in Subjects With Diabetic Gastroparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SP850
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2008-05

CONDITIONS: Diabetic Gastroparesis

INTERVENTIONS:
Drug: Reglan ODT

SUMMARY:
To determine whether a new Orally Disintegrating Tablet of Reglan (metoclopramide) is metabolized faster than the conventional Reglan tablet in patients with diabetic gastroparesis, pharmacokinetics following a single 10 mg dose of each formulation are being compared. Subjects must be 18 or older, have Type 1 or 2 diabetes with documented gastroparesis and agree to withhold medications for gastroparesis for 3 days prior to each dosing. Exclusion criteria include serum glucose >300 mg/dL, Hb1Ac >10%, and concurrent illness interfering with gastrointestinal motility. Subjects will stay in the clinic overnight, and pharmacokinetic sampling will continue for 8 hours after the first morning dose. The time (Tmax) and amount (Cmax) of peak concentration and the area under the curve (AUC) from time zero to 8 hr will be compared for the 2 formulations.

DETAILED DESCRIPTION:
See approved Package Insert for Adverse Event information.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 or older, have Type 1 or 2 diabetes with documented gastroparesis

Exclusion Criteria:

* Serum glucose >300 mg/dL, HbA1C >10%, and concurrent illness interfering with gastrointestinal motility

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-06; Primary Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Witt, Study Director — UCB Pharma
Locations (1):
- Schwarz, Milwaukee, Wisconsin, United States